CLINICAL TRIAL: NCT06542419
Title: The Effect of Selective Brain Cooling on Electrophysiological and Neuroinflammatory Biomarkers of Cognition and Mood
Brief Title: Brain Cooling Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Semyon M. Slobounov, Ph.D., Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Brain Cooling Biomarkers
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-08

CONDITIONS: Mental Health; Neurological Health
Keywords: Electroencephalography (EEG); Brain cooling; Neuroinflammation; Cytokines; Mental health; Depression; Anxiety
MeSH Terms: conditions — Psychological Well-Being; Neuroinflammatory Diseases; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This will be a straight forward parallel intervention model. Even numbers of participants will be randomly assigned to the treatment or control arms. The treatment group will receive the brain cooling intervention during their visits, while the control group will not. All other environmental, timing, and testing measures will remain constant between the groups as indicated in the study description.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brain Cooling Treatment (Experimental): Brain cooling consists of a 30-minute seated period, in a dimly lit, quiet room, while listening to calming natural sounds, during which they will wear an Arctic Cooling Cap V1.30, set at a temperature of 33.0 degrees Fahrenheit. Participants will be asked to remain awake, refrain from observing a screen, and relax to the best of their ability.
  This brain cooling treatment will occur on 7 consecutive days.
  Interventions: Device: Brain Cooling
- Control (No Intervention): The control arm consists of a 30-minute seated period, in a dimly lit, quiet room, while listening to calming natural sounds. Participants will be asked to remain awake, refrain from observing a screen, and relax to the best of their ability.

INTERVENTIONS:
Device: Brain Cooling — Brain cooling consists of a 30-minute seated period, in a dimly lit, quiet room, while listening to calming natural sounds, during which they will wear an Arctic Cooling Cap V1.30, set at a temperature of 33.0 degrees Fahrenheit. Participants will be asked to remain awake, refrain from observing a screen, and relax to the best of their ability. This brain cooling treatment will occur on 7 consecutive days.
  Other Names: Selective brain cooling; Cooling cap
  Arms: Brain Cooling Treatment

SUMMARY:
This research is being done to examine the effects of brain cooling on cognition, electrophysiological brain activity via EEG scans, inflammation of the brain, and mood in healthy subjects. Brain cooling has been shown to cause temporary symptom relief after traumatic brain injury, but its implications for general brain and mental health remain unexplored.

DETAILED DESCRIPTION:
This research attempts to address gaps in the current literature about the effect of selective brain cooling (SBC) on cognition, mood, electrophysiological markers of brain health and neuroinflammation in healthy subjects. In this study, the investigators will examine the short-term effect of one session of 30 minutes of brain cooling is on EEG patterns, neuroinflammation, cognition, and mood. The investigators will also examine the effect of a week-long intervention of 30 minutes of brain cooling per day on EEG patterns, neuroinflammation, cognition, mood. The overarching goal of this study is to validate the inclusion of selective brain cooling as an easy and safe addition to general health and clinical practice dedicated to cognitive and mood related neuropsychological health.

A minimum of 24 participants will be recruited for this study. 8 days of consecutive visits will be scheduled based on participant availability. Brain cooling consists of a 30-minute seated period, in a dimly lit, quiet room, while listening to calming natural sounds, during which the participants will wear an Arctic Cooling Cap V1.30, set at a temperature of 33.0 degrees Fahrenheit. Participants will be asked to remain awake, refrain from observing a screen, and relax in a wakeful state to the best of their ability. Participants assigned to the control group will be instructed similarly, but the brain cooling cap will not be functional.

The trial will consist of a 1-week daily intervention period and three major measurement time points: pre-intervention on Day 1, conclusion of Day 1, and post-intervention on Day 8. Day 1 will last approximately 105 minutes and will consist of 6 parts: completion of study consent form (10 min), saliva swab (5 min), administration of questionnaires and cognitive tests (10 min), electroencephalography (EEG) (20 mins), brain cooling or seated rest (30 mins), repeat questionnaires (10 mins), and repeat EEG (20 mins). The intervention period will consist of 7 days of daily administration of either 30 minutes of brain cooling or 30 minutes of seated rest. Day 8 will last approximately 35 minutes and will consist of: saliva swab (5 min), administration of questionnaires (10 min), electroencephalography (EEG) (20 mins).

Questionnaires administered to the participants at T1 and T2 will include: Penn State Worry Questionnaire (PSWQ), Hamilton Anxiety Rating Scale (HAM-A), Beck's Depression Inventory-Fast Screen (BDI-FS), Digit Span Test, Digit Symbol Test, Trail Making Test. All questionnaires and tests will be administered verbally or with paper and pencil.

Cheek swabs will be taken after the completion of the initial questionnaires. The process is as follows: for each subject the tester will use 10 swabs. Five swabs will be used to rub inside the left part of the mouth, and the other five will be used to rub inside the right part of the mouth. The exact area that will be swabbed will include the inside of the cheek, lip, and gums. This will be completed with a little pressure against the mouth and turning the swab slightly during the process. This will last approximately 20 seconds per swab. This cheek swab will allow us to test for levels of neuroinflammatory enzymes present in saliva.

EEG will be administered using a 19-channel EEG cap and analyzed using Neuroguide V2.8. Participants will be asked to maintain a seated position, while the EEG cap is fitted and proper electroconductance of all 19 electrodes is established with the scalp. This is done by injecting electroconduction gel through opening in each electrode using a blunt needle. Next, electrophysiological signal is recorded from the electrode cap for a 3-minute period. EEG in non-invasive and very minimal risk to the participant, with the exception of slight discomfort from adjustments to the cap on sensitive scalps or maintenance of the seated position for up to 20 minutes.

Brain cooling consists of a 30-minute seated period, in a dimly lit, quiet room, while listening to calming natural sounds, during which participants will wear an Arctic Cooling Cap V1.30, set at a temperature of 33.0 degrees Fahrenheit. Participants will be asked to remain awake, refrain from observing a screen, and relax to the best of their ability. Participants assigned to the control group will be instructed similarly, with the exclusion having the cooling cap turned on.

Directly following either the brain cooling or rest period, neuropsychological tests and questionnaires and EEG administration will be repeated prior to the subject leaving.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years old.

Exclusion Criteria:

* Not currently recovering from neurological injury or illness.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Trail Making Test | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  The Trail Making Test asks participants to trace a line connecting numbers and letters in logical order around a page. They are timed. It tests cognition and processing speed.
Digit Span Test | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  The Digit Span test ask participants to repeat strings of digits in either normal or reverse order to test cognition and working memory.
Beck's Depression Inventory-Fast Screen | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  The Beck's Depression Inventory-Fast Screen is a 13-item subjective report of depression symptoms.
HAM-A | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  the HAM-A is a 14-item subjective report of anxiety symptoms.
Digit Symbol Test | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  The Digit Symbol Test is a 90 second test that requires subjects to continually match numbers 1-9 with corresponding symbols. This test measures processing speed, inhibition, and general cognition.
Neuroinflammatory Cytokines | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  We will use the saliva acquired from cheek swabs to assess degree of circulating neuroinflammatory serum biomarkers. Specifically, we will examine the cytokines CRP and IL-6 which have been shown to be associated with neurological trauma and brain health.
The Penn State Worry Questionnaire | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  The Penn State Worry Questionnaire is a 16-item subjective report of perceived worry.
EEG Pattern | The metrics will be assessed pre-intervention (beginning of Day 1), after the acute effect of brain cooling (at the end of Day 1), and after the chronic effect of brain cooling (Day 8).
  The investigators will use the data acquired from EEG to measure specific electrophysiological metrics (electrical field potential from brain activity). Specifically, we will isolate whole-brain relative alpha-power and relative beta-power.

CONTACTS AND LOCATIONS:
Locations (1):
- Recreation Building, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walter A, Finelli K, Bai X, Johnson B, Neuberger T, Seidenberg P, Bream T, Hallett M, Slobounov S. Neurobiological effect of selective brain cooling after concussive injury. Brain Imaging Behav. 2018 Jun;12(3):891-900. doi: 10.1007/s11682-017-9755-2. PMID 28712093
- [Background] Tan XR, Stephenson MC, Alhadad SB, Loh KWZ, Soong TW, Lee JKW, Low ICC. Elevated brain temperature under severe heat exposure impairs cortical motor activity and executive function. J Sport Health Sci. 2024 Mar;13(2):233-244. doi: 10.1016/j.jshs.2023.09.001. Epub 2023 Sep 9. PMID 37678507
- [Background] Westermaier T, Nickl R, Koehler S, Fricke P, Stetter C, Rueckriegel SM, Ernestus RI. Selective Brain Cooling after Traumatic Brain Injury: Effects of Three Different Cooling Methods-Case Report. J Neurol Surg A Cent Eur Neurosurg. 2017 Jul;78(4):397-402. doi: 10.1055/s-0036-1596057. Epub 2016 Dec 30. PMID 28038481
- [Background] Leung LY, Cardiff K, Yang X, Srambical Wilfred B, Gilsdorf J, Shear D. Selective Brain Cooling Reduces Motor Deficits Induced by Combined Traumatic Brain Injury, Hypoxemia and Hemorrhagic Shock. Front Neurol. 2018 Aug 3;9:612. doi: 10.3389/fneur.2018.00612. eCollection 2018. PMID 30123177
- [Background] Deng H, Han HS, Cheng D, Sun GH, Yenari MA. Mild hypothermia inhibits inflammation after experimental stroke and brain inflammation. Stroke. 2003 Oct;34(10):2495-501. doi: 10.1161/01.STR.0000091269.67384.E7. Epub 2003 Sep 11. PMID 12970518
- [Background] undefined
- [Background] Congeni J, Murray T, Kline P, Bouhenni R, Morgan D, Liebig C, Lesak A, McNinch NL. Preliminary Safety and Efficacy of Head and Neck Cooling Therapy After Concussion in Adolescent Athletes: A Randomized Pilot Trial. Clin J Sport Med. 2022 Jul 1;32(4):341-347. doi: 10.1097/JSM.0000000000000916. Epub 2021 Mar 10. PMID 34009790
- See also: publication from the Journal of Cerebral Blood Flow Metabolism describing use of this product in the methods — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9580175/
- See also: Aspen Cooling Systems (product designer) — https://aspensystems.com/system-applications/medical/cold-caps/